CLINICAL TRIAL: NCT02410850
Title: Long Term Oral Appliance Therapy Effectiveness for Obstructive Sleep Apnea: A Multicenter Cohort Study
Brief Title: Long Term Oral Appliance Therapy Effectiveness for Obstructive Sleep Apnea Syndrome
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Universiteit Antwerpen (Other); University of Sydney (Other); University Hospital, Angers (Other Government); University of Groningen (Other); Université de Montréal (Other); Kaiser Permanente (Other); Stanford University (Other); Laval University (Other); University of Cambridge (Other); Kyushu University (Other); Japan Somnology Center, Neuropsychiatric Research Institute (Unknown); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fernanda Almeida, Principle Investigator, University of British Columbia
Other Study IDs: H14-00743
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral Appliance; objective adherence; cardiovascular events; cardiovascular mortality; cerebrovascular mortality; cost effectiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (13):
- University of Montreal: Patients from University of Montreal in Canada
  Interventions: Device: Oral Appliance
- University of Antwerp: Patients from University of Antwerp in Belgium.
  Interventions: Device: Oral Appliance
- University of Sydney: Patients from University of Sydney in Australia.
  Interventions: Device: Oral Appliance
- Angers University Hospital: Patients from Angers University Hospital in France.
  Interventions: Device: Oral Appliance
- University of Gronigen: Patients from University of Gronigen in Netherlands.
  Interventions: Device: Oral Appliance
- Kaiser Permanente: Patients from Kaiser Permanente from USA.
  Interventions: Device: Oral Appliance
- Stanford University: Patients from Stanford University from USA.
  Interventions: Device: Oral Appliance
- Laval University: Patients from Laval University in Canada.
  Interventions: Device: Oral Appliance
- Cambridge University: Patients from Cambridge University in UK.
  Interventions: Device: Oral Appliance
- Kyushu University: Patients from Kyushu University in Japan
  Interventions: Device: Oral Appliance
- Japan Somnology Center: Patients from Japan Somnology Center in Japan.
  Interventions: Device: Oral Appliance
- Uniformed Services University: Patients from the Uniformed Services University in USA.
  Interventions: Device: Oral Appliance
- University of British Columbia: Patients from the University of British Columbia in Canada.
  Interventions: Device: Oral Appliance

INTERVENTIONS:
Device: Oral Appliance — Mandibular Advancement Splints

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent breathing problem that occurs during sleep. OSA have been associated with the obesity epidemic in developing countries; additionally, high OSA prevalence rates are present in populations with cardiovascular and metabolic disorders. Two OSA treatments are currently available, oral appliance (OA) therapy and continuous positive airway pressure (CPAP). OAs are an underutilized non-surgical treatment and few studies have analyzed their long-term effectiveness for patients with OSA. The purpose of this study is to assess the long-term effectiveness of OA therapy in patients with OSA and to explore any changes on cardiovascular related morbidity and mortality related to this therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a chronic condition which may occur when an individual is sleeping. OSA incidence rates ranges from 4 to 16% of the adult population. The prevalence of OSA is even higher in populations with cardiovascular and metabolic disorders (e.g. stroke or diabetes mellitus).

OSA is characterized by five or more pauses in breathing per hour or partial obstruction of airway during sleep.

Obstructive sleep apnea (OSA) is currently being treated using two methods: oral appliance (OA) therapy and continuous positive airway pressure (CPAP). Although the American Academy of Sleep Medicine (AASM) has approved both methods as a first line treatment for mild and moderate OSA, oral appliances have been underutilized despite their non-invasive, quietness, the fact they are non-surgical and, cost effectiveness. OAs can also be an alternative for severe OSA patients who find CPAP treatment intolerable. There are two major groups of OAs available, one that acts on repositioning the mandible and tongue; this includes mandibular advancement splints (MAS) and Mandibular advancement devices (MAD). The other group of OAs, tongue retaining devices (TRD) focus on holding the tongue forward. It is because of the positioning of the tongue and mandible that OAs is effective in decreasing sleep apnea. OA therapy is a long-term treatment and therefore it is important that the appliance be comfortable to encourage patient use.

Despite the benefits to patients using OAs, previous studies have not looked at the relationship between OAs and OSA in long term studies or in a large number of patients. This lack of research and knowledge has led to an absence in training and education for dentists who are able to provide OA therapy to their patients. OAs have been shown to not be as effective as CPAP in helping with OSA, however, it has similar effects on blood pressure, quality of life, sleepiness and endothelial function. Previous studies have shown that the effects of OA therapy on patients' OSA are associated with more acceptance and adherence. Previous longitudinal studies that followed patients using CPAP showed great benefits in terms of cardiovascular health. It is therefore necessary for large sample size, long term prospective cohort studies to be done to determine how effective OA therapy is for patients with OSA, while also looking at potential effects on cardiovascular morbidity and mortality. It is for this reason that 15 centres from 9 counties around the world have formed a network called ORANGE (Oral Appliance Network on Global Effectiveness) dedicated on the long-term outcomes of OAs.

These centers included: University of Sidney (Australia), Stanford University (USA). Kaiser Permanente (USA), Cambridge University (UK), Paris Hospital (France), University of Antwerp (Belgium), Japan Somnology Center (Japan), Kyushu University (Japan), University of British Columbia (Canada), University of Montreal (Canada), Laval University (Canada), University of Gronigen (Netherlands), and Umea University (Sweden).

ELIGIBILITY:
Inclusion Criteria:

* Patients are currently prescribed Oral Appliance for their Obstructive Sleep Apnea

Exclusion Criteria:

* Patients under the age of 18 years.
* Patients that do not understand the English language.
* Patients that refuse to sign the informed consent for any reason.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who seek Oral Appliance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Long term effectiveness of Oral Appliance therapy by assessing responses to treatment specific questionnaires and other questionnaires such as Functional Outcomes of Sleep Questionnaire (FOSQ), Epworth Sleepiness Scale(ESS), and Short Form 36 (SF-36) | 5 years
Impact of Oral Appliance therapy on cardiovascular morbidity by assessing health changes, hospitalizations and number of deaths during treatment with Oral Appliance | 5 years
Impact of Oral Appliance therapy on cardiovascular mortality by assessing health changes, hospitalizations and number of deaths during treatment with Oral Appliance | 5 years

SECONDARY OUTCOMES:
Objective adherence by assessing Oral Appliance adherence chip data | 1,3,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Almeida, DDS,Phd, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada